CLINICAL TRIAL: NCT01967940
Title: A Phase 3, Two-Part Study to Evaluate the Efficacy of Tenofovir Alafenamide Versus Placebo Added to a Failing Regimen Followed by Treatment With Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Plus Atazanavir in HIV-1 Positive, Antiretroviral Treatment-Experienced Adults
Brief Title: Efficacy of Tenofovir Alafenamide Versus Placebo Added to a Failing Regimen Followed by Treatment With Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Plus Atazanavir in HIV-1 Positive, Antiretroviral Treatment-Experienced Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-292-0117; 2013-002830-19 (EudraCT Number)
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-07

CONDITIONS: HIV; HIV Infections; Acquired Immunodeficiency Syndrome
Keywords: HIV-1; HIV; Treatment-Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — tenofovir alafenamide; Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Atazanavir Sulfate

STUDY DESIGN:
Intervention Model Description: Part 1 (Sentinel Cohort followed by a Randomized Cohort), 14-day washout period, then Part 2
Who Masked: Participant, Investigator
Masking Description: Part 1 Sentinel Cohort: Open-label, non-randomized Part 1 Randomized Cohort: Double-blind, randomized Part 2: Open-label, non-randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 Sentinel Cohort (TAF) (Experimental): TAF + their current failing ARV regimen for 10 days in Part 1
  Interventions: Drug: TAF; Drug: Current failing ARV regimen
- Part 1 Randomized Cohort (TAF) (Experimental): Following review of safety and efficacy data from the Sentinel Cohort, participants will be randomized to receive TAF + their current failing ARV regimen for 10 days in Part 1.
  Interventions: Drug: TAF; Drug: Current failing ARV regimen
- Part 1 Randomized Cohort (Placebo) (Placebo Comparator): Following review of safety and efficacy data from the Sentinel Cohort, participants will be randomized to receive placebo + their current failing ARV regimen for 10 days in Part 1.
  Interventions: Drug: Placebo; Drug: Current failing ARV regimen
- Part 2 E/C/F/TAF+ATV (Experimental): Following a 14-day period to confirm eligibility, participants in the Randomized Cohort TAF group with a > 0.5 log10 decline in HIV-1 RNA and all participants completing the Randomized Cohort Placebo group will receive E/C/F/TAF+ATV for 48 weeks in Part 2. After completion of Part 2, all participants will be eligible to continue to receive E/C/F/TAF plus ATV in the extension phase until E/C/F/TAF becomes commercially available, or until Gilead Sciences terminates development of E/C/F/TAF in the applicable country.
  Interventions: Drug: E/C/F/TAF; Drug: ATV

INTERVENTIONS:
Drug: TAF — 25 mg tablet administered orally once daily with food
  Other Names: Vemlidy®; GS-7340
  Arms: Part 1 Randomized Cohort (TAF); Part 1 Sentinel Cohort (TAF)
Drug: Placebo — Tablets to match TAF administered orally once daily with food
  Arms: Part 1 Randomized Cohort (Placebo)
Drug: E/C/F/TAF — 150/150/200/10 mg STR administered orally once daily with food
  Other Names: Genvoya®
  Arms: Part 2 E/C/F/TAF+ATV
Drug: Current failing ARV regimen — Participants will continue taking their current ARV regimen as prescribed in Part 1.
  Arms: Part 1 Randomized Cohort (Placebo); Part 1 Randomized Cohort (TAF); Part 1 Sentinel Cohort (TAF)
Drug: ATV — 300 mg tablet administered orally once daily.
  Other Names: Reyataz®
  Arms: Part 2 E/C/F/TAF+ATV

SUMMARY:
The primary objective of this study is to evaluate the efficacy of tenofovir alafenamide (TAF) versus placebo, each administered with the existing, failing antiretroviral (ARV) regimen. There are 2 parts to this study: Part 1 and Part 2.

Part 1 consists of 2 cohorts, starting with a sentinel cohort, in which participants will be enrolled to receive open-label TAF in addition to their current failing ARV regimen. This cohort will then be followed by a randomized, double-blind, cohort to compare the addition of TAF or placebo in HIV-1 positive adults who are failing their current ARV regimen.

In Part 2, all participants who complete Part 1 of the study will discontinue their failing ARV regimen and TAF or placebo for a 14-day washout period. Following the washout period, all participants who received TAF in Part 1 and have a > 0.5 log10 decline in HIV-1 RNA will receive elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) single-tablet regimen (STR) plus atazanavir (ATV) once daily for 48 weeks. Participants who received TAF who have a ≤ 0.5 log10 decline in HIV-1 RNA will be discontinued from the study and will not be eligible to continue into Part 2 of the study. All participants who received placebo in Part 1 will be eligible to participate in Part 2 regardless of their viral load change. After completion of Part 2, all participants will be eligible to continue to receive E/C/F/TAF plus ATV in the extension phase until E/C/F/TAF becomes commercially available, or until Gilead Sciences terminates development of E/C/F/TAF in the applicable country.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* Currently taking a failing ARV regimen
* Plasma HIV-1 RNA ≥ 500 copies/mL but ≤ 100,000 copies/mL at screening
* Normal ECG
* Estimated glomerular filtration rate (eGFR) ≥ 50 mL/min according to the Cockcroft-Gault formula for creatinine clearance
* Alanine aminotransferase (AST)/aspartate aminotransferase (AST) ≤ 5 × the upper limit of the normal range (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function
* Serum amylase ≤ 5 × ULN
* Females may enter the study if it is confirmed that she is:

  * Not pregnant or nursing
  * Of non-childbearing potential (ie, have had a hysterectomy, both ovaries removed, medically documented ovarian failure, or are postmenopausal women > 54 years of age with cessation [for ≥ 12 months] of previously occurring menses), or
  * Of childbearing potential and agrees to utilize highly effective contraception methods or be non-heterosexually active or practice sexual abstinence from screening throughout the duration of study treatment and for 30 days following study drug dosing

    * Females who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing.
* Males must agree to utilize a highly effective method of contraception during heterosexual intercourse or be non-heterosexually active, or practice sexual abstinence from first dose throughout the study period and for 30 days following the last study drug dose.
* Males must agree to refrain from sperm donation from first dose until at least 30 days after the last study drug dose.

Key Exclusion Criteria:

* A new AIDS-defining condition diagnosed within the 30 days prior to screening
* Hepatitis B surface antigen (HBsAg) positive
* Hepatitis C antibody positive (individuals with positive hepatitis C virus (HCV) antibody and without detectable HCV RNA are permitted to enroll)
* History of integrase inhibitor use
* Screening or historical genotype reports shows Q151M or T69ins or more than 3 TAMs.
* Screening or historical genotype report shows resistance to integrase inhibitors
* Individuals experiencing decompensated cirrhosis
* Current alcohol or substance use
* History of malignancy within the past 5 years (prior to screening) or ongoing malignancy other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma, or resected, non-invasive cutaneous squamous carcinoma. Individuals with cutaneous KS are eligible, but must not have received any systemic therapy for KS within 30 days of Part 1, Day 1 and must not be anticipated to require systemic therapy during the study.
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to Part 1, Day 1
* Any other clinical condition or prior therapy that would make the individual unsuitable for the study or unable to comply with dosing requirements
* Participation in any other clinical trial (including observational trials) without prior approval from the sponsor is prohibited while participating in this trial
* Receiving ongoing therapy with any disallowed medications, including any drugs not to be used with elvitegravir, cobicistat, emtricitabine and tenofovir alafenamide or known allergies to the excipients of E/C/F/TAF STR

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-10-25 (Actual); Primary Completion 2015-05-21 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (15):
- United States (5):
  - Midway Immunology and Research center, Ft. Pierce, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Rowan Tree Medical, P.A., Wilton Manors, Florida
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
- Dominican Republic (2):
  - Salvador B Gautier Hospital - Infectious Diseases Department, Santo Domingo
  - Instituto Dominicano de Estudio Virologicos - IDEV, Santo Domingo
- Russia (2):
  - Regional state budget health agency Krasnoyarsk Regional Center for Prevention and Control of AIDS, Krasnoyarsk
  - Center For Prevention and Treatment of AIDS and Infectious Diseases, Saint Petersburg, Saint Petersburg
- Thailand (5):
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Bangkok
  - Ramathibodi Hospital, Mahidol University, Bangkok
  - Siriraj Hospital Department of Preventive and Social Medicine, Faculty of Medicine, Bangkok
  - Chiang Mai University, Chiang Mai
  - Khon Kaen University, Khon Kaen
- Joint Clinical Research Centre, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Uganda, Thailand, Russian Federation, and Dominican Republic. The first participant was screened on 25 October 2013. The last study visit occurred on 31 July 2017.
Pre-assignment Details: 259 participants were screened.
Groups:
- Part 1 Sentinel Cohort TAF: Tenofovir alafenamide (TAF) 25 mg tablet once daily + their current failing regimen for 10 days
- Part 1 Randomized Cohort TAF: TAF 25 mg tablet once daily + their current failing regimen for 10 days
- Part 1 Randomized Cohort Placebo: Placebo once daily + their current failing regimen for 10 days
- Part 2 E/C/F/TAF + ATV: Following a 14 day washout period, participants from the Randomized Cohort TAF group who had a > 0.5 log10 decline in HIV-1 RNA and participants from the Randomized Cohort Placebo group were eligible to receive elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) (150/150/200/10 mg) single-tablet regimen (STR) plus atazanavir (ATV) 300 mg once daily for 48 weeks. After completion of Part 2, all participants were eligible to continue to receive E/C/F/TAF plus ATV in the extension phase until E/C/F/TAF became commercially available, or until Gilead Sciences terminated development of E/C/F/TAF in the applicable country.
Period: Part 1
Arm/Group | Part 1 Sentinel Cohort TAF | Part 1 Randomized Cohort TAF | Part 1 Randomized Cohort Placebo | Part 2 E/C/F/TAF + ATV
Started | 12 | 28 | 15 | 0
Completed | 12 | 28 | 15 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1 Sentinel Cohort TAF | Part 1 Randomized Cohort TAF | Part 1 Randomized Cohort Placebo | Part 2 E/C/F/TAF + ATV
Started | 0 (4 participants completed Part 1 and did not enter Part 2; 8 participants moved to the Part 2 group) | 0 (12 participants completed Part 1 and did not enter Part 2; 16 participants moved to the Part 2 group) | 0 (1 participant completed Part 1 and did not enter Part 2; 14 participants moved to the Part 2 group) | 38 (38 participants from the Part 1 groups moved to this Part 2 E/C/F/TAF + ATV group)
Completed | 0 | 0 | 0 | 35
Not Completed | 0 | 0 | 0 | 3
Not completed — Enrolled in Part 2 and Never Treated | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Unknown Reason | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: participants who enrolled into Part 1 of the study and received at least one dose of study drug in Part 1.
Groups:
- Part 1 Sentinel Cohort TAF; Part 1 Randomized Cohort TAF: TAF 25 mg tablet once daily + their current failing regimen for 10 days
- Total: Total of all reporting groups
Arm/Group | Part 1 Sentinel Cohort TAF | Part 1 Randomized Cohort TAF | Part 1 Randomized Cohort Placebo | Total
Number analyzed (Participants) | 12 | 28 | 15 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (7.3) | 40 (9.1) | 43 (8.2) | 40 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 16 | 4 | 23
  Male | 9 | 12 | 11 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 1 | 6
  Not Hispanic or Latino | 7 | 28 | 14 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 5 | 5 | 10
  Black | 3 | 22 | 9 | 34
  White | 4 | 1 | 0 | 5
  Other | 5 | 0 | 1 | 6
Region of Enrollment [Number; unit: participants]
  Russian Federation | 2 | 1 | 0 | 3
  United States | 5 | 3 | 0 | 8
  Dominican Republic | 5 | 0 | 1 | 6
  Uganda | 0 | 19 | 9 | 28
  Thailand | 0 | 5 | 5 | 10
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.18 (0.648) | 4.16 (0.544) | 4.03 (0.953) | 4.13 (0.688)
HIV-1 RNA Category [Count of Participants; unit: Participants]
  ≤ 100,000 copies/mL | 12 | 27 | 12 | 51
  > 100,000 to ≤ 400,000 copies/mL | 0 | 1 | 3 | 4
CD4 Cell Count [Mean (Standard Deviation); unit: cells/µL] | 269 (207.1) | 245 (244.6) | 232 (162.4) | 246 (213.7)
CD4 Percentage [Mean (Standard Deviation); unit: percentage] | 17.4 (10.14) | 16.5 (11.09) | 14.3 (8.61) | 16.1 (10.15)

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants With Plasma HIV-1 RNA Decreases From Baseline Exceeding 0.5 log10 at Day 10
Time Frame: Day 10
Population: Part 1 Full Analysis Set: participants who enrolled into Part 1 of the study and received at least one dose of study drug in Part 1.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Sentinel Cohort TAF | Part 1 Randomized Cohort TAF | Part 1 Randomized Cohort Placebo
Number analyzed (Participants) | 12 | 28 | 15
percentage of participants | 58.3 | 60.7 | 0
Statistical Analysis 1: Comparison: Part 1 Randomized Cohort TAF vs Part 1 Randomized Cohort Placebo; A sample size of 90 participants, randomized in a 2:1 ratio, achieves 89% power to detect a 35% difference in the proportion of participants with HIV-1 RNA decreases from baseline exceeding 0.5 log10 between the TAF and placebo arms at Day 10. Sample size and power computation was based on the assumption that 50% of participants in the TAF arm and 15% of participants in the placebo arm achieved a reduction exceeding 0.5 log10 HIV-1 RNA; Test type: Superiority — Enrollment into this study was stopped early due to the challenge of recruiting a sufficient number of participants who met the eligibility criteria. The actual number of enrolled is 55, among them 43 enrolled in the Randomized Cohort. Based on the actual enrollment numbers, the power to detect a 35% difference drops to 51%, under the same assumptions in the original sample size calculations; p < 0.001, Fisher Exact; Difference in proportions = 60.7, 95% CI 2-sided [42.6 to 78.8] — The 95% confidence interval was estimated based on unconditional exact method using 2 inverted 1-sided tests with the standardized statistic

2. Secondary Outcome: Part 1: Change From Baseline in Plasma log10 HIV-1 RNA (Copies/mL) at Day 10
Time Frame: Baseline; Day 10
Population: Part 1 Full Analysis Set
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Part 1 Sentinel Cohort TAF | Part 1 Randomized Cohort TAF | Part 1 Randomized Cohort Placebo
Number analyzed (Participants) | 12 | 28 | 15
log10 copies/mL | -0.72 (0.574) | -0.70 (0.628) | -0.04 (0.233)

3. Secondary Outcome: Part 2: Safety of E/C/F/TAF STR Plus ATV in Participants Who Switched From a Failing Regimen as Assessed by the Percentage of Participants Experiencing Grade 3 or 4 Laboratory Abnormalities Through Week 24
Time Frame: Up to Week 24
Population: Part 2 Safety Analysis Set: participants who enrolled into Part 2 of the study and received at least one dose of study drug in Part 2.
Measure: Number; unit: percentage of participants
Groups:
- Part 2 E/C/F/TAF + ATV: E/C/F/TAF (150/150/200/10 mg) STR plus ATV 300 mg once daily for 48 weeks
Arm/Group | Part 2 E/C/F/TAF + ATV
Number analyzed (Participants) | 37
percentage of participants | 37.8

4. Secondary Outcome: Part 2: Safety of E/C/F/TAF STR Plus ATV in Participants Who Switched From a Failing Regimen as Assessed by the Percentage of Participants Experiencing Grade 3 or 4 Laboratory Abnormalities Through Week 48
Time Frame: Up to Week 48
Population: Part 2 Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 E/C/F/TAF + ATV
Number analyzed (Participants) | 37
percentage of participants | 48.6

5. Secondary Outcome: Part 2: Safety of E/C/F/TAF STR Plus ATV in Participants Who Switched From a Failing Regimen as Assessed by the Percentage of Participants Experiencing Any Treatment-Emergent Adverse Event Through Week 24
Time Frame: Up to Week 24
Population: Part 2 Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 E/C/F/TAF + ATV
Number analyzed (Participants) | 37
percentage of participants | 75.7

6. Secondary Outcome: Part 2: Safety of E/C/F/TAF STR Plus ATV in Participants Who Switched From a Failing Regimen as Assessed by the Percentage of Participants Experiencing Any Treatment-Emergent Adverse Event Through Week 48
Time Frame: Up to Week 48
Population: Part 2 Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 E/C/F/TAF + ATV
Number analyzed (Participants) | 37
percentage of participants | 81.1

7. Secondary Outcome: Part 2: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL as Defined by the FDA Snapshot Analysis at Week 24
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: Part 2 Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 E/C/F/TAF + ATV
Number analyzed (Participants) | 37
percentage of participants | 86.5

8. Secondary Outcome: Part 2: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL as Defined by the FDA Snapshot Analysis at Week 48
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Part 2 Full Analysis Set: participants who enrolled into Part 2 of the study and received at least one dose of study drug in Part 2.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 E/C/F/TAF + ATV
Number analyzed (Participants) | 37
percentage of participants | 97.3

9. Secondary Outcome: Part 2: Percentage of Participants With Plasma HIV-1 RNA < 400 Copies/mL as Defined by the FDA Snapshot Analysis at Week 24
Description: The percentage of participants with HIV-1 RNA < 400 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: Part 2 Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 E/C/F/TAF + ATV
Number analyzed (Participants) | 37
percentage of participants | 94.6

10. Secondary Outcome: Part 2: Percentage of Participants With Plasma HIV-1 RNA < 400 Copies/mL as Defined by the FDA Snapshot Analysis at Week 48
Description: The percentage of participants with HIV-1 RNA < 400 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Part 2 Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 E/C/F/TAF + ATV
Number analyzed (Participants) | 37
percentage of participants | 97.3

11. Secondary Outcome: Part 2: Change From Baseline in Plasma log10 HIV-1 RNA (Copies/mL) at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the Part 2 Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Part 2 E/C/F/TAF + ATV
Number analyzed (Participants) | 35
log10 copies/mL | -2.96 (0.754)

12. Secondary Outcome: Part 2: Change From Baseline in Plasma log10 HIV-1 RNA (Copies/mL) at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Part 2 Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Part 2 E/C/F/TAF + ATV
Number analyzed (Participants) | 35
log10 copies/mL | -3.04 (0.594)

13. Secondary Outcome: Part 2: Change From Baseline in CD4+ Cell Count at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the Part 2 Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Part 2 E/C/F/TAF + ATV
Number analyzed (Participants) | 35
cells/μL | 76 (92.8)

14. Secondary Outcome: Part 2: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Part 2 Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Part 2 E/C/F/TAF + ATV
Number analyzed (Participants) | 35
cells/μL | 125 (109.0)

15. Secondary Outcome: Part 2: Change From Baseline in CD4+ Percentage at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the Part 2 Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Part 2 E/C/F/TAF + ATV
Number analyzed (Participants) | 35
percentage change | 4.4 (2.35)

16. Secondary Outcome: Part 2: Change From Baseline in CD4+ Percentage at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Part 2 Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Part 2 E/C/F/TAF + ATV
Number analyzed (Participants) | 35
percentage change | 5.7 (2.99)

ADVERSE EVENTS:
Time Frame: Baseline up to the last dose date plus 30 days (average exposure: Part 1 = 10 days; Part 2 = 86.5 weeks)
Description: Safety Analysis Set: participants who enrolled into the study and received at least one dose of study drug.
Groups:
- Part 2 E/C/F/TAF + ATV: E/C/F/TAF (150/150/200/10 mg) STR plus ATV 300 mg once daily for 48 weeks plus the extension phase
Arm/Group | Part 1 Sentinel Cohort TAF | Part 1 Randomized Cohort TAF | Part 1 Randomized Cohort Placebo | Part 2 E/C/F/TAF + ATV
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/28 | 0/15 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/12 | 3/28 | 0/15 | 4/37
Other Adverse Events (participants affected / at risk) | 7/12 | 6/28 | 5/15 | 26/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Sentinel Cohort TAF (N=12) | Part 1 Randomized Cohort TAF (N=28) | Part 1 Randomized Cohort Placebo (N=15) | Part 2 E/C/F/TAF + ATV (N=37)
Enlarged uvula (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Sentinel Cohort TAF (N=12) | Part 1 Randomized Cohort TAF (N=28) | Part 1 Randomized Cohort Placebo (N=15) | Part 2 E/C/F/TAF + ATV (N=37)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Chest pain (General disorders) | 0 | 0 | 0 | 2
Malaise (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 3
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 3
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 1 | 0 | 3
Malaria (Infections and infestations) | 0 | 0 | 0 | 5
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 1
Pyuria (Infections and infestations) | 0 | 0 | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 11
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 2
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 4
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Eosinophilic cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years